CLINICAL TRIAL: NCT07386314
Title: Motor and Cognitive Telerehabilitation for Acquired Brain Injury
Acronym: TELEGCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Toscana Nord Ovest (Other)
Collaborators: IRCCS Bonino Pulejo (Unknown); Istituto S.Anna Crotone (Unknown)
Responsible Party: Principal Investigator, Federico Posteraro, Head of rehabilitation department Versilia Hospital, Azienda USL Toscana Nord Ovest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUSL Toscana Nord Ovest
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Acquired Brain Injury
Keywords: Brain Injury; tele-rehabilitation; motor; cognitive
MeSH Terms: conditions — Brain Injuries | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Presence (GP) (Experimental): Patients in the in-person treatment group (GP) will undergo 50-minute sessions, three times a week, for a total of eight weeks using VRRS virtual reality systems (Khymeia, Padua, Italy), certified Class A medical devices.
  Interventions: Device: Group Presence
- Group Tele-Rehabilitation (Active Comparator): The telerehabilitation treatment group (GT) will receive a similar motor and cognitive treatment program at home using the VRRS HomeKit device (Khymeia, Padua, Italy), another certified Class 1 medical device.
  Interventions: Device: Tele-rehabilitation

INTERVENTIONS:
Device: Tele-rehabilitation — The telerehabilitation treatment group (GT) will receive a similar motor and cognitive treatment program at home using the VRRS HomeKit device (Khymeia, Padua, Italy), another certified Class 1 medical device.
  Arms: Group Tele-Rehabilitation
Device: Group Presence — Patients in the in-person treatment group (GP) will undergo 50-minute sessions, three times a week, for a total of eight weeks using VRRS virtual reality systems (Khymeia, Padua, Italy), certified Class 1 medical devices. The first four weeks of treatment will be conducted with VRRS EVO, while the following four weeks will be conducted with VRRS Physio, with exercises designed to improve various cognitive and motor domains of the upper limb.
  Arms: Group Presence (GP)

SUMMARY:
The overall objective of the study is to compare upper limb cognitive and motor rehabilitation programs delivered via tele-rehabilitation and in-person, in order to evaluate their overall impact on the rehabilitation process of subjects with GCA outcomes at the end of the subacute phase.

DETAILED DESCRIPTION:
The study is a controlled clinical trial aimed at evaluating the efficacy and feasibility of cognitive and motor rehabilitation programs delivered in person or via tele-rehabilitation. Sixty-two subjects, aged 18 to 75, of both sexes, will be consecutively enrolled at the three participating centers. The sample size was calculated assuming a change of 15 points (standard deviation 20) on the Brief Neuropsychological Examination (BNE), with alpha = 0.05, beta = 0.2, and a power of 80%. A 10% margin was added to the resulting number (28 subjects per group) for potential dropouts. The ENB was chosen as the primary measure because, validated in the Italian population, it allows for a comprehensive, multidomain assessment that is sensitive to changes in the main cognitive domains (attention, memory, language, executive and praxic functions), also allowing for the evaluation of treatment efficacy over time, with short administration times and good tolerability in patients with GCA outcomes. Recent multicenter studies have confirmed its reliability and clinical relevance in this population. Subjects will be assigned to two treatment groups using block randomization, stratified by age, gender, and baseline functional level. This procedure was adopted to reduce potential bias and ensure greater comparability between groups. However, a geographical restriction will be maintained: patients unable to physically access the facility will be included in the tele-rehabilitation group (TG), but will follow the same stratification and randomization procedure, ensuring methodological consistency and allowing for dedicated sensitivity analyses.

The in-person treatment group (GP) will complete 50-minute sessions, three times a week for eight weeks, at the rehabilitation center. The tele-rehabilitation treatment group (TG) will complete a similar program at home, with the same frequency and duration, via dedicated platforms.

Sixty-two subjects (18-75 years old, both genders) will be consecutively enrolled at the three participating centers upon discharge from hospital rehabilitation. Patients will be assigned equally to the two groups (in-person treatment and tele-rehabilitation) using block randomization stratified by age, gender, and functional level.

ELIGIBILITY:
Inclusion Criteria:

Outcome of Severe Acquired Brain Injury (GAI) of various etiologies;

* Age between 18 and 75 years
* Level of Cognitive Functioning (LCF) at discharge from the hospital ward >= 6;
* One or more neuropsychological deficits in the areas of attention, memory, language, and executive functions;
* Possible upper limb motor deficit;
* Absence of general clinical complications that could interfere with rehabilitation treatment;
* Cognitive and language functions sufficient to understand the instructions provided and give consent -

Exclusion Criteria:

* Level of Cognitive Functioning (LCF) at discharge from hospitalization ward < 6;
* Presence of previous deficits in neuropsychological and motor functions prior to the acute event;
* Vulnerable subjects or those in emergency situations
* Failure to provide informed consent.
* Pregnant or intending to become pregnant during the enrollment period -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Brief Neuropshychological Examination | Pre-intervetion and immediately after 8 weeks of intervention
Flug Meyer Upper Extremity Scale | Pre-intervetion and immediately after 8 weeks of intervention

SECONDARY OUTCOMES:
System Usability Scale | Pre-intervetion and immediately after 8 weeks of intervention
Client Satisfaction Questionnaire-8 Total scores range from 8 to 32, with the higher number indicating greater satisfaction | Pre-intervetion and immediately after 8 weeks of intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maggio MG, Rizzo A, De Francesco M, Barbera M, Kamran M, De Luca R, Corallo F, Quartarone A, Calabro RS. What About the Differences in Body Representation and Body Image Between Stroke Patients and Healthy Controls? Psychological and Clinical Implications. Brain Behav. 2025 May;15(5):e70155. doi: 10.1002/brb3.70155. PMID 40342223
- [Background] Maggio MG, Bonanno L, Rizzo A, Barbera M, Benenati A, Impellizzeri F, Corallo F, De Luca R, Quartarone A, Calabro RS. The role of virtual reality-based cognitive training in enhancing motivation and cognitive functions in individuals with chronic stroke. Sci Rep. 2025 Jul 12;15(1):25258. doi: 10.1038/s41598-025-08173-1. PMID 40652006
- [Background] De Luca R, Calderone A, Gangemi A, Rifici C, Bonanno M, Maggio MG, Cappadona I, Veneziani I, Ielo A, Corallo F, Quartarone A, Cardile D, Calabro RS. Is Virtual Reality Orientation Therapy Useful to Optimize Cognitive and Behavioral Functioning Following Severe Acquired Brain Injury? An Exploratory Study. Brain Sci. 2024 Apr 23;14(5):410. doi: 10.3390/brainsci14050410. PMID 38790389
- See also: Related Info — https://simfer.it/consensus-conference-cicerone-documento-finale-conclusivo/